CLINICAL TRIAL: NCT02198872
Title: Effects of Aquatic and Land Aerobic Training on Body Composition and Cardiorespiratory and Metabolic Variables in Patients With Cardiorespiratory Diseases
Brief Title: Aquatic and Land Aerobic Training, Cardiorespiratory and Metabolic Variables in Cardiorespiratory Diseases
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Universidade Metodista de Piracicaba (Other)
Responsible Party: Principal Investigator, Elie Fiogbé, Professor, Universidade Metodista de Piracicaba
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 03/13; 190729/2011-2 (Other Grant/Funding Number: 190729/2011-2)
Record Dates: First submitted 2014-07-15; First posted 2014-07-24 (Estimated); Last update posted 2014-07-24 (Estimated); Status verified 2014-07

CONDITIONS: Arteriosclerosis, Coronary
Keywords: Autonomic Nervous System, Body composition, Oxygen Uptake,; Water Based Physical Training, Land Based Physical Training.
MeSH Terms: conditions — Coronary Artery Disease | interventions — Exercise

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Exercise, Aerobic (Water based) (Experimental): Patients of this group will be submitted to an aerobic water based physical training
  Interventions: Other: Exercise, Aerobic (Water based)
- Land Group (Active Comparator): Patients of this group perform physical training on bicycle.
  Interventions: Other: Land Group

INTERVENTIONS:
Other: Exercise, Aerobic (Water based) — Patients of this group will be submitted to an aerobic water based physical training
  Arms: Exercise, Aerobic (Water based)
Other: Land Group — Patients of this group perform physical training on bicycle.
  Arms: Land Group

SUMMARY:
In the pathophysiological process of coronary artery disease (CAD), are present, autonomic dysfunction and reduced functional capacity. Studies showed that physical training (PT) is critical in the treatment of CAD by promoting beneficial effects. Although water based exercises program have been documented in patients with various cardiovascular diseases, the most of studies among patients with CAD used land based exercises programs. OBJECTIVE: To evaluate and compare the effects of aerobic water (WPT) and land (LPT) based PT on autonomic modulation of heart rate (HR), body composition and cardiorespiratory and metabolic variables in patients with CAD. METHODS : 40 men between 50 and 70 years old with CAD diagnosed by coronary angiography showing obstruction greater than 50% and underwent angioplasty will be evaluated in 4 stages; 1) immediately after angioplasty, clinical assessment, body composition analysis and recording of HR and NN intervals during rest. 2) The components of step 1) will be repeated after three month, adding the record of HR and NN before, during and after the Valsalva maneuver, spirometry and cardiopulmonary exercise testing. 3) Volunteers will be randomly divided into two groups, WPT and LPT for 48 sessions. 4) The components of step 2) are repeated after each period of 12 sessions. Thus, it is expected that WPT promote beneficial physiological adaptations in CAD patients with obstruction greater than 50%.

DETAILED DESCRIPTION:
1. Immediately after angioplasty, the volunteers will be subject to an assessment (Assessment 0), which will consist of:

   * History: personal data, lifestyle and food, family history, current and previous history of disease.
   * Physical examination: cardiac and lung auscultation,measurement of heart rate (HR), blood pressure (BP), body weight and height.
   * Analysis of body composition by bioelectrical impedance analysis.
   * Registration of HR and NN intervals (NN) during rest, in the supine and sitting positions.
   * biochemical blood tests: complete blood count, blood glucose, total cholesterol, LDL and HDL cholesterol, triglycerides, and C-reactive protein ultrasensitive.
   * Recording of HR and NN during rest in the supine position, sitting, standing and during respiratory sinus arrhythmia maneuver.
2. Three months after the "Assessment 0", the volunteers will be subject to an assessment (initial Assessment) prior to physical training program. Will be repeated all assessments performed in the "Assessment 0" plus the record of HR and R-Ri before, during and after the Valsalva maneuver, spirometry and cardiopulmonary exercise test (CPET). This is a submaximal CPET performed on a treadmill, in order to verify and identify possible changes in hemodynamic, electrocardiographic induced to physical exertion, their aerobic functional capacity as well as to prescribe physical training protocol.
3. After this assessment, the volunteers will be randomly assigned to one of two groups, aerobic water (WPT) or land (LPT) based physical training.
4. Components of "Initial Assessment" will be repeated at the end of each month of physical training (Revaluation 1, 2 and 3) and the end (Final Assessment).

ELIGIBILITY:
Inclusion Criteria:

* diagnosis by angiography
* sedentaries
* family story of cardiac disease
* obesity

Exclusion Criteria:

* frequent arrhythmias at rest
* triggered by physical effort
* unstable angina
* chronic obstructive pulmonary disease
* insulin-dependent diabet
* renal failure
* sequel of stroke
* uncontrolled hypothyroidism
* water phobia
* skin infections, allergic reactions to chlorine,
* urinary incontinence and
* musculoskeletal and neuromuscular disorders precluding physical tests and training sessions

Ages: 50 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2014-09; Primary Completion 2015-07 (Estimated); Study Completion 2018-02 (Estimated)

PRIMARY OUTCOMES:
Change in autonomic system modulation | baseline and 16 weeks
  Change in autonomic system modulation in assess by comparing the heart rate variability at baseline and after a 16 weeks of aerobic water and land based physical training.

SECONDARY OUTCOMES:
Change in body composition | 16 weeks
  Change in body composition is assess by comparing the body composition at baseline and after a 16 weeks of aerobic water and land based physical training.

OTHER OUTCOMES:
Oxygen uptake | 16 Weeks
  Change in oxygen uptake is assessed by comparing the oxygen uptake at baseline and after a 16 weeks of aerobic water and land based physical training.

CONTACTS AND LOCATIONS:
Overall Officials: Elie Fiogbé, Ms, Principal Investigator — Universidade Metodista de Piracicaba
Locations (1):
- Universidade Metodista de Piracicaba, Piracicaba, São Paulo, Brazil